CLINICAL TRIAL: NCT05590117
Title: The Possible Protective Effect of Pentoxifylline Against Chemotherapy Induced Toxicities in Patients With Colorectal Cancer
Brief Title: Protective Effect of Pentoxifylline Against Chemotherapy Induced Toxicities in Patients With Colorectal Cancer
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Tarek Aboelnoor, Principal Investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 35931/10/22
Record Dates: First submitted 2022-10-13; First posted 2022-10-21 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Colo-rectal Cancer; Neuropathy;Peripheral; Mucositis
Keywords: Colorectal cancer; Neuropathy; Mucositis; Pentoxifylline; Chemotherapy; Toxicity
MeSH Terms: conditions — Colonic Neoplasms; Neuritis; Mucositis; Colorectal Neoplasms | interventions — Pentoxifylline; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 placebo (Placebo Comparator): n=24 which will receive 12 cycles of FOLFOX-6 regimen plus placebo tablets twice daily.
  Interventions: Drug: Placebo; Drug: FOLFOX-6 regimen
- Group 2 pentoxifylline (Active Comparator): n=24 which will receive FOLFOX-6 regimen in addition to pentoxifylline 400 mg twice daily.
  Interventions: Drug: Pentoxifylline; Drug: FOLFOX-6 regimen

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline is a potent anti inflammatory may prevent chemotherapy induced neuropathy and mucositis and will be administered 400mg twice daily
  Other Names: Trental
  Arms: Group 2 pentoxifylline
Drug: Placebo — placebo tablets
  Arms: Group 1 placebo
Drug: FOLFOX-6 regimen — 12 cycles of FOLFOX-6 regimen
  Other Names: Oxaliplatin, Fluorouracil, calcium leucovorin

SUMMARY:
This study aims to:

- Evaluate the possible protective effect of pentoxifylline against oxaliplatin induced peripheral neuropathy and chemotherapy induced mucositis in patients with stage II and stage III colorectal cancer.

This study will be a randomized placebo controlled parallel study.48 patients with colorectal cancer will be randomized to 2 groups:

Group I (control group; n=24) which will receive 12 cycles of FOLFOX-6 regimen plus placebo tablets twice daily. Group II (Pentoxiphylline group; n=24) which will receive FOLFOX-6 regimen in addition to pentoxifylline 400 mg twice daily.

Blood sample collection and biochemical assessment:

* Malondialdehyde (MDA) as oxidative stress marker (colorimetry).
* Tumor necrosis factor alfa (TNF-α) as pro inflammatory marker (ELISA).
* Neurotensin (NT) as a potential marker for neuropathic pain (ELISA).
* Citrulline as a biomarker for mucositis (ELISA).

Clinical assessment of oxaliplatin induced neuropathy will be done through:

The assessment of the severity of neuropathic pain through "Brief Pain Inventory-Short Form" at baseline and by the end of every two chemotherapy cycles.

The implication of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, Version 5, 2017) for grading of neuropathy every 2 cycles. The use of Neurotoxicity- 12 item questionnaire score (Ntx-12) from the validated Functional Assessment of Cancer Therapy/Gynecologic Oncology Group at baseline and by the end of every two chemotherapy cycles).

Mucositis will be assessed at baseline and by the end of every two chemotherapy cycles through the use of common terminology criteria for adverse events "CTCAE, version 5.00, 2017

DETAILED DESCRIPTION:
This study aims to:

- Evaluate the possible protective effect of pentoxifylline against oxaliplatin induced peripheral neuropathy and chemotherapy induced mucositis in patients with stage II and stage III colorectal cancer.

This study will be a randomized placebo controlled parallel study.48 patients with colorectal cancer will be randomized to 2 groups:

Group I (control group; n=24) which will receive 12 cycles of FOLFOX-6 regimen plus placebo tablets twice daily. Group II (Pentoxiphylline group; n=24) which will receive FOLFOX-6 regimen in addition to pentoxifylline 400 mg twice daily.

Blood sample collection and biochemical assessment:

* Malondialdehyde (MDA) as oxidative stress marker (colorimetry).
* Tumor necrosis factor alfa (TNF-α) as pro inflammatory marker (ELISA).
* Neurotensin (NT) as a potential marker for neuropathic pain (ELISA).
* Citrulline as a biomarker for mucositis (ELISA).

Clinical assessment of oxaliplatin induced neuropathy will be done through:

The assessment of the severity of neuropathic pain through "Brief Pain Inventory-Short Form" at baseline and by the end of every two chemotherapy cycles.

The implication of National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE, Version 5, 2017) for grading of neuropathy every 2 cycles. The use of Neurotoxicity- 12 item questionnaire score (Ntx-12) from the validated Functional Assessment of Cancer Therapy/Gynecologic Oncology Group at baseline and by the end of every two chemotherapy cycles).

Mucositis will be assessed at baseline and by the end of every two chemotherapy cycles through the use of common terminology criteria for adverse events "CTCAE, version 5.00, 2017. Assessment of participants' adherence, side effects and tolerability Pentoxiphylline will be provided on biweekly basis and the participants' adherence will be assessed through counting the returned tablets. Participants will be followed-up by weekly telephone calls and direct meetings during chemotherapy cycles to assess their adherence and to report any drug related adverse effects. The adverse effects will be collected and graded according to the National Cancer Institute Common Terminology Criteria for Adverse events "NCI-CTCAE; version 5, 2017". Participants will be considered non- adherent and excluded from the study if not consumed the provided tablets or lost the follow-up meeting at any time of intervention or changed regimen.

The primary and secondary endpoints:

The primary endpoint is the percentage of patients with peripheral sensory neuropathy grade ≥ 2, the variation of 12-item neurotoxicity questionnaire (Ntx- 12) total score and the variation in grades of mucositis. The secondary endpoint is the change in the serum concentrations of the measured biological markers.

Sample size calculation:

According to the results of previous studies, the total number of subjects required to detect the effect of neuro-protective drugs in patients received neuro- toxic chemotherapy was 41 patients with 5% significance, 80% statistical power and an attrition of 15 %. In this context, during the current study, a total sample size of 41 patients in both arms will be sufficient to detect the effect. Assuming that the attrition rate will be 15 %, the initial sample size will be 48 patients in both arms with 24 patients in each arm.

Ethical approval:

The study will be performed in accordance with the ethical standards of Helsinki declaration in 1964 and its later amendments. The study will be approved by the Research Ethics Committee of Tanta University. The study will be registered as a clinical trial at ClinicalTrials.gov. All participants will be informed about the benefits and risks of the study. Any unexpected risks that will appear during the course of the research will be clarified to the participants and to the ethical committee on time. The data of the enrolled patients will be confidential. All enrolled patients will give their written informed consents. The study will be conducted between October 2022 and October 2024.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with histologically confirmed diagnosis of stage II and stage III colorectal cancer.
* Patients who will be scheduled to receive FOLFOX-6 regimen.
* Patients with no contraindication to chemotherapy.
* Males and females aged ≥ 18 years old.
* Adequate baseline hematologic values (absolute neutrophilic count ≥ 1.5

  × 109/L, platelet count ≥ 100 × 109/L and hemoglobin level ≥ 10 g/dl).
* Patients with adequate renal function (serum creatinine < 1.5 mg/dL and Creatinine clearance (ClCr) ˃ 45 mL/min).
* Patients with adequate liver function (serum bilirubin < 1.5 mg/dl).
* Patients with performance status < 2 according to Eastern Cooperative Oncology Group (ECOG) score.

Exclusion Criteria:

* - Children < 18 years old.
* Prior exposure to neurotoxic chemotherapy (oxaliplatin, cisplatin, vincristine, paclitaxel, docetaxel or Isoniazid) for at least 6 months prior the study treatment.
* Evidence of pre-existing peripheral neuropathy resulting from another reason (diabetes, brain tumor or brain trauma).
* Patients with diabetes and other conditions that predispose to neuropathy as hypothyroidism, autoimmune diseases or hepatitis C.
* History of known allergy to oxaliplatin or other platinum agents.
* Patients with other inflammatory diseases (rheumatoid arthritis and ulcerative colitis) or stressful conditions (obesity class 2 and 3, smoking).
* Concomitant use of multivitamins (vitamins E, C and A), tricyclic antidepressants or other neuro-protective medications (gabapentin, lamotrigine, carbamazepine and phenytoin, etc...).
* Concurrent active cancer originating from a primary site other than colon or rectum.
* Patients on blood thinning agents
* Pregnant and breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-10-11 (Estimated); Primary Completion 2023-10-11 (Estimated); Study Completion 2024-10-11 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with peripheral sensory neuropathy grade ≥ 2 | 6 months
  Grading according to National Cancer Institute Common Terminology. there are 5 grades; Grade (1) is asymptomatic may be accompanied by loss of tendon reflex or paresthesia. Grade (2) is moderate symptoms which limit instrumental activities of daily life Grade (3) is severe symptoms which limit self-care activates of daily life. Grade (4) is life threatening consequences or urgent intervention indicated. Grade (5) is death.
  Criteria for Adverse Events (NCI-CTCAE, Version 5, 2017)
variation of 12-item neurotoxicity questionnaire (Ntx- 12) total score | 6 months
  the Ntx-12 questionnaire is comprised of 12 statements intended to measure the severity and impact of peripheral sensory neuropathy on patients' lives. Patients will be instructed to complete the Arabic version of the Ntx-12 and choose the number corresponding to how true each statement was for them using a likert-type scale, with 0 indicating not at all; 1, a little bit; 2, somewhat; 3, quite a bit; and 4, very much
variation in grades of mucositis | 6 months
  Mucositis will be assessed through the use of common terminology criteria for adverse events "CTCAE, version 5.00, 2017". Grade (1) is Asymptomatic or mild symptoms; intervention not indicated. Grade (2) is Moderate pain or ulcer that does not interfere with oral intake; modified diet indicated. Grade (3) is Severe pain, interfering with oral intake. Grade (4) is Life-threatening consequences; urgent intervention indicated. Grade (5) is Death.

SECONDARY OUTCOMES:
Change in the biological marker Malondialdehyde | 6 months
  Malondialdehyde (MDA) as oxidative stress marker will be measured using colorimetry
Change in the biological marker Tumor necrosis factor alfa | 6 months
  Tumor necrosis factor alfa (TNF-α) as pro inflammatory marker will be measured using ELISA will be measured using (ELISA).
Change in the biological marker Neurotensin | 6 months
  Neurotensin (NT) as a potential marker for neuropathic pain will be measured using ELISA
Change in the biological marker Citrulline | 6 months
  Citrulline as a biomarker for mucositis will be measured using ELISA

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbyia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keum N, Giovannucci E. Global burden of colorectal cancer: emerging trends, risk factors and prevention strategies. Nat Rev Gastroenterol Hepatol. 2019 Dec;16(12):713-732. doi: 10.1038/s41575-019-0189-8. Epub 2019 Aug 27. PMID 31455888
- [Background] Guren MG. The global challenge of colorectal cancer. Lancet Gastroenterol Hepatol. 2019 Dec;4(12):894-895. doi: 10.1016/S2468-1253(19)30329-2. Epub 2019 Oct 21. No abstract available. PMID 31648973
- [Background] Andre T, Iveson T, Labianca R, Meyerhardt JA, Souglakos I, Yoshino T, Paul J, Sobrero A, Taieb J, Shields AF, Ohtsu A, Grothey A, Sargent DJ; for the IDEA Steering Committee. The IDEA (International Duration Evaluation of Adjuvant Chemotherapy) Collaboration: Prospective Combined Analysis of Phase III Trials Investigating Duration of Adjuvant Therapy with the FOLFOX (FOLFOX4 or Modified FOLFOX6) or XELOX (3 versus 6 months) Regimen for Patients with Stage III Colon Cancer: Trial Design and Current Status. Curr Colorectal Cancer Rep. 2013;9(3):261-269. doi: 10.1007/s11888-013-0181-6. PMID 24032000
- [Background] Zedan AH, Hansen TF, Fex Svenningsen A, Vilholm OJ. Oxaliplatin-induced neuropathy in colorectal cancer: many questions with few answers. Clin Colorectal Cancer. 2014 Jun;13(2):73-80. doi: 10.1016/j.clcc.2013.11.004. Epub 2013 Nov 13. PMID 24365057
- [Background] Saito Y, Okamoto K, Kobayashi M, Narumi K, Furugen A, Yamada T, Iseki K. Magnesium co-administration decreases cisplatin-induced nephrotoxicity in the multiple cisplatin administration. Life Sci. 2017 Nov 15;189:18-22. doi: 10.1016/j.lfs.2017.08.028. Epub 2017 Aug 31. PMID 28864226
- [Background] Hoff PM, Saad ED, Costa F, Coutinho AK, Caponero R, Prolla G, Gansl RC. Literature review and practical aspects on the management of oxaliplatin-associated toxicity. Clin Colorectal Cancer. 2012 Jun;11(2):93-100. doi: 10.1016/j.clcc.2011.10.004. Epub 2011 Dec 6. PMID 22154408
- [Background] Zanardelli M, Micheli L, Cinci L, Failli P, Ghelardini C, Di Cesare Mannelli L. Oxaliplatin neurotoxicity involves peroxisome alterations. PPARgamma agonism as preventive pharmacological approach. PLoS One. 2014 Jul 18;9(7):e102758. doi: 10.1371/journal.pone.0102758. eCollection 2014. PMID 25036594
- [Background] Chakraborty A, Chowdhury S, Bhattacharyya M. Effect of metformin on oxidative stress, nitrosative stress and inflammatory biomarkers in type 2 diabetes patients. Diabetes Res Clin Pract. 2011 Jul;93(1):56-62. doi: 10.1016/j.diabres.2010.11.030. Epub 2010 Dec 13. PMID 21146883
- [Background] Kleczkowska P, Lipkowski AW. Neurotensin and neurotensin receptors: characteristic, structure-activity relationship and pain modulation--a review. Eur J Pharmacol. 2013 Sep 15;716(1-3):54-60. doi: 10.1016/j.ejphar.2013.03.004. Epub 2013 Mar 14. PMID 23500196
- [Background] Plaza-Manzano G, Molina-Ortega F, Lomas-Vega R, Martinez-Amat A, Achalandabaso A, Hita-Contreras F. Changes in biochemical markers of pain perception and stress response after spinal manipulation. J Orthop Sports Phys Ther. 2014 Apr;44(4):231-9. doi: 10.2519/jospt.2014.4996. Epub 2014 Jan 22. PMID 24450367
- [Background] Al Moundhri MS, Al-Salam S, Al Mahrouqee A, Beegam S, Ali BH. The effect of curcumin on oxaliplatin and cisplatin neurotoxicity in rats: some behavioral, biochemical, and histopathological studies. J Med Toxicol. 2013 Mar;9(1):25-33. doi: 10.1007/s13181-012-0239-x. PMID 22648527
- [Background] Basile D, Di Nardo P, Corvaja C, Garattini SK, Pelizzari G, Lisanti C, Bortot L, Da Ros L, Bartoletti M, Borghi M, Gerratana L, Lombardi D, Puglisi F. Mucosal Injury during Anti-Cancer Treatment: From Pathobiology to Bedside. Cancers (Basel). 2019 Jun 20;11(6):857. doi: 10.3390/cancers11060857. PMID 31226812
- [Background] Fragkos KC, Forbes A. Citrulline as a marker of intestinal function and absorption in clinical settings: A systematic review and meta-analysis. United European Gastroenterol J. 2018 Mar;6(2):181-191. doi: 10.1177/2050640617737632. Epub 2017 Oct 12. PMID 29511548
- [Background] Yehia R, Saleh S, El Abhar H, Saad AS, Schaalan M. L-Carnosine protects against Oxaliplatin-induced peripheral neuropathy in colorectal cancer patients: A perspective on targeting Nrf-2 and NF-kappaB pathways. Toxicol Appl Pharmacol. 2019 Feb 15;365:41-50. doi: 10.1016/j.taap.2018.12.015. Epub 2018 Dec 25. PMID 30592963
- [Background] Speer EM, Dowling DJ, Ozog LS, Xu J, Yang J, Kennady G, Levy O. Pentoxifylline inhibits TLR- and inflammasome-mediated in vitro inflammatory cytokine production in human blood with greater efficacy and potency in newborns. Pediatr Res. 2017 May;81(5):806-816. doi: 10.1038/pr.2017.6. Epub 2017 Jan 10. PMID 28072760
- [Background] Tan G, Jensen MP, Thornby JI, Shanti BF. Validation of the Brief Pain Inventory for chronic nonmalignant pain. J Pain. 2004 Mar;5(2):133-7. doi: 10.1016/j.jpain.2003.12.005. PMID 15042521
- [Background] Freites-Martinez A, Santana N, Arias-Santiago S, Viera A. Using the Common Terminology Criteria for Adverse Events (CTCAE - Version 5.0) to Evaluate the Severity of Adverse Events of Anticancer Therapies. Actas Dermosifiliogr (Engl Ed). 2021 Jan;112(1):90-92. doi: 10.1016/j.ad.2019.05.009. Epub 2020 Sep 3. No abstract available. English, Spanish. PMID 32891586
- [Background] Kidwell KM, Yothers G, Ganz PA, Land SR, Ko CY, Cecchini RS, Kopec JA, Wolmark N. Long-term neurotoxicity effects of oxaliplatin added to fluorouracil and leucovorin as adjuvant therapy for colon cancer: results from National Surgical Adjuvant Breast and Bowel Project trials C-07 and LTS-01. Cancer. 2012 Nov 15;118(22):5614-22. doi: 10.1002/cncr.27593. Epub 2012 May 8. PMID 22569841
- [Background] Vondracek P, Oslejskova H, Kepak T, Mazanek P, Sterba J, Rysava M, Gal P. Efficacy of pregabalin in neuropathic pain in paediatric oncological patients. Eur J Paediatr Neurol. 2009 Jul;13(4):332-6. doi: 10.1016/j.ejpn.2008.06.011. Epub 2008 Sep 6. PMID 18774740
- [Background] Salehifar E, Janbabaei G, Hendouei N, Alipour A, Tabrizi N, Avan R. Comparison of the Efficacy and Safety of Pregabalin and Duloxetine in Taxane-Induced Sensory Neuropathy: A Randomized Controlled Trial. Clin Drug Investig. 2020 Mar;40(3):249-257. doi: 10.1007/s40261-019-00882-6. PMID 31925721

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT05590117/Prot_SAP_000.pdf